CLINICAL TRIAL: NCT03284567
Title: A Randomized Controlled Trial to Investigate the Health Promoting Effects of a Football Fitness Intervention for Women After Treatment for Breast Cancer
Brief Title: Football Fitness After Breast Cancer
Acronym: FFABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jacob Uth, Postdoc, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FFABC
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Breast Neoplasm Female
Keywords: Breast cancer; Football; Late effects; Physical exercise; Soccer training; Rehabilitation; Bone mineralization; Body composition; Fitness; Aerobic capacity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: 1/3 of participants will be randomly allocated to the control group and 2/3 of participants will be randomly allocated to the Football fitness intervention group.
Who Masked: Outcomes Assessor
Masking Description: Personnel assessing the primary outcome is blinded for study participants group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Football fitness (Active Comparator): Participants in the intervention group will practice soccer for 52 weeks two times weekly. A soccer instructor will be in charge of all training sessions. The training will consist of 30 min of warm-up exercises (running, dribbling, passing, shooting, balance and muscle strength exercises), followed by 2 x 15 minutes of 4-7 a-side games.
  Training will take place on a natural grass pitch. In adverse weather conditions (i.e., < 5°C or heavy rain) training will be performed indoors. Participants will be told to avoid hard tackles and other actions that carry a risk of injury.
  Interventions: Behavioral: Football fitness
- Control group (No Intervention): Participants in the control group will receive verbal advice about the benefits of exercise and physical activity.

INTERVENTIONS:
Behavioral: Football fitness — The training will consist of 30 min of warm-up exercises (running, dribbling, passing, shooting, balance and muscle strength exercises), followed by 2 x 15 minutes of 4-7 a-side games.
  Training will take place on a natural grass pitch. In adverse weather conditions (i.e., < 5°C or heavy rain) training will be performed indoors
  Arms: Football fitness

SUMMARY:
Late effects of breast cancer treatment are widely reported including deteriorating fitness, fatigue, loss of muscle and bone mass, and increased body fat percentage. Exercise interventions may ameliorate a number of these effects including fatigue, fitness and improve quality of life. However only limited knowledge exists on the potential of novel interventions and settings, such as sports outside the hospital setting, to improve late effects of breast cancer treatment. The 'Football Fitness After Breast Cancer' (FF ABC) study is a randomized trial comparing the effects of a football training intervention with standard treatment approaches on fitness, bone mineralization, body composition, muscle strength, blood pressure, and patient-reported outcomes in women treated for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women surgically managed for breast cancer, local and regional advanced breast cancer.
* Completion of adjuvant chemotherapy and radiation therapy.
* Legally competent persons with ability to read and understand Danish.
* Signed informed consent.
* Performance level 0-1 (WHO).

Exclusion Criteria:

* WHO performance level > 1.
* Osteoporosis (T-score < -2.5).
* Known metastatic breast cancer (stage IV).
* Women in DBCG-group I (age => 60 years, tumor =< 10 mm, invasive ductal carcinoma grade I, invasive lobular carcinoma grade I / II, estrogen receptor positive and HER2 normal).
* Cardiovascular or pulmonary disorders (e.g., arrhythmias, ischemic heart disease, unregulated high blood pressure, chronic obstructive lung disease).
* Ongoing anticoagulant therapy (vitamin K antagonists; Marevan, Marcoumar and low molecular weight heparins; Innohep, Clexane, Fragmin) for pulmonary embolism or deep venous thrombosis (DVT) due to increased bleeding risk of falls and clashes with other players during exercise.
* Current or scheduled chemotherapy and radiation therapy in the intervention period (12 months).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Mean change in fitness level (maximal oxygen uptake) from baseline to month 6 and month 12. | 6 months and 12 months.
  Incremental test to exhaustion on a cycle ergometer.

SECONDARY OUTCOMES:
Mean change in whole-body fat mass from baseline to month 6 and month 12. | 6 months and 12 months.
  Assessed by dual energy x-ray absorptiometry.
Mean change in whole-body weight from baseline to month 6 and month 12. | 6 month and 12 month.
  Body weight was measured with a digital platform scale.
Mean change in whole-body muscle mass from baseline to month 6 and month 12. | 6 month and 12 month.
  Assessed by dual energy x-ray absorptiometry.
Mean change in muscle strength from baseline to month 6 and month 12. | 6 month and 12 month.
  Dynamic concentric muscle strength for the knee extensors (1RM).
Mean change in balance from baseline to month 6 and month 12. | 6 month and 12 month.
  Single-leg flamingo balance test.
Mean change in blood pressure from baseline to month 6 and month 12. | 6 month and 12 month.
  Blood pressure will be measured with a digital sphygmomanometer.
Mean change in markers of bone mineral metabolism from baseline to month 6 and month 12. | 6 month and 12 month.
  Procollagen type I C propeptide, osteocalcin and C-terminal telopeptide will be analyzed by a chemiluminescence method using a fully automated immunoassay system (iSYS, Immunodiagnostic Systems Ltd., Boldon, England.
Mean change in cholesterol from baseline to month 6 and month 12. | 6 month and 12 month.
  Blood samples will be analyzed at baseline, 6 and 12 month for total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglycerides, and glycosylated hemoglobin, respectively, by automated analyzers (Cobas Fara, Roche, Neuilly sur Seine, France) using enzymatic kits (Roche Diagnostics, Mannheim, Germany, and Tosoh G7, Tosoh Europe, Tessenderlo, Belgium).
Self-reported physical activity from baseline to month 6 and month 12. | 6 month and 12 month.
  Assessed by the International Physical Activity Questionnaire (IPAQ).
Self-reported diagnosis-specific symptoms and side-effects from baseline to month 6 and month 12. | 6 month and 12 month.
  Assessed by the supplement EORTC QLQ-BR23.
Self-reported health-related quality of life outcomes from baseline to month 6 and month 12. | 6 month and 12 month.
  Assessed by the 15 subscales of the European Organization for Research and Treatment of Cancer (EORTC QLQ-C30).
Self-reported functional level in upper extremities from baseline to month 6 and month 12. | 6 month and 12 month.
  Assessed by disabilities of the arm, shoulder and hand (DASH).
Self-reported health related quality of life from baseline to month 6 and month 12. | 6 month and 12 month.
  Assessed by The Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36)
Mean change in bone mineral density (BMD) of the spine (L2-L4), Total hip and Femoral Neck. | 6 month and 12 month.
  Assessed by dual energy x-ray absorptiometry.
Mean change in total body and leg bone mineral content (BMC). | 6 month and 12 month.
  Assessed by dual energy x-ray absorptiometry.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Copenhagen, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bloomquist K, Krustrup P, Fristrup B, Sorensen V, Helge JW, Helge EW, Soelberg Vadstrup E, Rorth M, Hayes SC, Uth J. Effects of football fitness training on lymphedema and upper-extremity function in women after treatment for breast cancer: a randomized trial. Acta Oncol. 2021 Mar;60(3):392-400. doi: 10.1080/0284186X.2020.1868570. Epub 2021 Jan 11. PMID 33423594
- [Derived] Uth J, Fristrup B, Sorensen V, Helge EW, Christensen MK, Kjaergaard JB, Moller TK, Mohr M, Helge JW, Jorgensen NR, Rorth M, Vadstrup ES, Krustrup P. Exercise intensity and cardiovascular health outcomes after 12 months of football fitness training in women treated for stage I-III breast cancer: Results from the football fitness After Breast Cancer (ABC) randomized controlled trial. Prog Cardiovasc Dis. 2020 Nov-Dec;63(6):792-799. doi: 10.1016/j.pcad.2020.08.002. Epub 2020 Aug 12. PMID 32800792